CLINICAL TRIAL: NCT01541059
Title: Postoperative Analgesia in Third Molar Surgery Under General Anesthesia: Ropivacaine Versus Placebo
Brief Title: Postoperative Analgesia Following Wisdom Teeth Removal: Ropivacaine Versus Placebo
Acronym: RopiMol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LOCAL/2011/JR/HG-02; 2011-004972-13 (EudraCT Number)
Record Dates: First submitted 2012-02-20; First posted 2012-02-29 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-10

CONDITIONS: Third Molar Extraction
Keywords: Third molar extraction; local anesthesia; ropivacaine
MeSH Terms: interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients in this arm will have standard anesthesia with the injection of placebo solution into the vestibular of each tooth to be extracted
  Interventions: Drug: Placebo injection
- Ropivacaine (Experimental): Patients in this arm will have general anesthesia with injection of ropivacaine into the vestibular next to each tooth to be extracted.
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Placebo injection — Injection of saline solution into the vestibular capsule of each tooth to be extracted.
  Other Names: Standard intervention; Saline solution
  Arms: Placebo
Drug: Ropivacaine injection — Ropivacaine is injected into the vestibular capsule of each tooth to be extracted.
  Other Names: Experimental intervention.
  Arms: Ropivacaine

SUMMARY:
The main objective of this study is to demonstrate the superiority of local analgesia with ropivacaine versus placebo on postoperative pain during the first 24 hours following bilateral surgery of all four third molars under general anesthesia.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare regional anesthesia by ropivacaine versus placebo for the bilateral resection of all four third molars under general anesthesia, in terms of:

A. intraoperative use of propofol and remifentanil B. postoperative pain (EVN) at different time points C. in-hospital analgesic consumption D. time to first rescue analgesic request E. time spent in the post interventional treatment room F. length of hospital stay G. side effects H. analgesic consumption at home I. analgesic consumption (total) J. patient satisfaction K. Chronic pain after surgery

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 3 months of follow-up
* American Society of Anesthesiology (ASA) score of 1, 2 or 3
* Patient programmed for surgical removal of all 4 wisdom teeth, excluding all other teeth, under general anesthesia

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is over 18 years old and under judicial protection, under tutorship or curatorship
* The patient (or legal representative)refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* Ineffective contraceptive
* Addiction or chronic pain treated with morphine
* Contra-indication for regional anesthesia (eg congenital or acquired coagulopathy, infection, allergy)
* Contra-indication to local anesthetics, general anesthetics and analgesics used in the protocol.
* Difficult cooperation, psychiatric disorders that could interfere with assessments
* Hypersensitivity to ropivacaine or other local anesthetics with amide links
* Contra-indication for the use of NaCl 0.9%: all states of sodium and water retention (especially heart failure, edema and ascites syndrome associated with cirrhosis)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08-29 (Actual); Study Completion 2015-08-29 (Actual)

PRIMARY OUTCOMES:
24 hour area under the curve for pain | 24 hours
  Pain is assessed via a numeric, verbal scale (0 to 10) at baseline and then at 1.5, 2, 3, 4, 6 and 24 hours after surgery. The area under the resulting curve is calculated.

SECONDARY OUTCOMES:
Total peroperative consumption of remifentanil | During surgery (approximately 30-50 minutes)
  µg/kg
Total peroperative consumption of propofol | During surgery (approximately 30-50 minutes)
  mg/kg
Post operative pain as measured by a verbal, numeric scale (0 to 10) | Day 1
  score from 0 to 10
Post operative pain as measured by a verbal, numeric scale (0 to 10) | Day 4
  score from 0 to 10
Post operative pain as measured by a verbal, numeric scale (0 to 10) | 1 month
  score from 0 to 10
Post operative pain as measured by a verbal, numeric scale (0 to 10) | 3 months
  score from 0 to 10
Total morphine consumption | Hospital discharge (on average on days 1 or 2)
  mg
Use of rescue pain medicine (yes/no) | Hospital discharge (on average on days 1 or 2)
Total in-hospital Tramadol consumption | Hospital discharge (on average on days 1 or 2)
  mg
Total in-hospital paracetamol consumption | Hospital discharge (on average on days 1 or 2)
  g
Total in-hospital ketoprofen consumption | Hospital discharge (on average on days 1 or 2)
  mg
Time elapsed between release from post-surgical recovery room and first request for rescue medicine | Hospital discharge (on average on days 1 or 2)
  minutes
Length of recovery room stay | Recovery room discharge (Day 1)
  Time elapsed between admittance and discharge from the post-surgical recovery room. (minutes)
Length of hospital stay | Hospital discharge (on average on days 1 or 2)
  Time elapsed between admittance to post-surgical recovery room and hospital discharge (hours)
presence/absence of complications | 6 hours
  pruritus, nausea, vomiting, bleeding, anesthesia of the mouth, difficulty breathing, drowsiness, headache, sweating, palpitations, skin rash, difficult glutition, dysarthria
presence/absence of complications | day 1
  pruritus, nausea, vomiting, bleeding, anesthesia of the mouth, difficulty breathing, drowsiness, headache, sweating, palpitations, skin rash, difficult glutition, dysarthria
presence/absence of complications | day 3
  pruritus, nausea, vomiting, bleeding, anesthesia of the mouth, difficulty breathing, drowsiness, headache, sweating, palpitations, skin rash, difficult glutition, dysarthria
Paracetamol consumption at home | Day 1
  grams
Paracetamol consumption at home | Day 3
  grams
ketoprofen consumption at home | Day 1
  mg
ketoprofen consumption at home | Day 3
  mg
Tramadol consumption at home | Day 1
  mg
Tramadol consumption at home | Day 3
  mg
Patient satisfaction | Day 3
  Patient satisfaction is evaluated via a numeric verbal scale ranging from 0 to 10.
Chronic pain evaluation (DN4) | 1 month
  standard DN4 score
Chronic pain evaluation (DN4) | 3 months
  standard DN4 score

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ripart, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France

REFERENCES:
- [Result] Ghezal H, Bouvet S, Kabani S, Ripart J, Cuvillon P. Ropivacaine versus placebo on postoperative analgesia and chronic pain following third molar extraction: A Prospective Randomized Controlled Study. J Stomatol Oral Maxillofac Surg. 2020 Apr;121(2):113-117. doi: 10.1016/j.jormas.2019.07.005. Epub 2019 Jul 18. PMID 31326593